CLINICAL TRIAL: NCT00187733
Title: Influence of OCTN2 Variants on Carnitine Status and Plasma Triglycerides
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 1005
Record Dates: First submitted 2005-09-14; First posted 2005-09-16 (Estimated); Last update posted 2012-09-13 (Estimated); Status verified 2012-09

CONDITIONS: Carnitine Transporter Deficiency
Keywords: L-carnitine
MeSH Terms: conditions — Systemic carnitine deficiency | interventions — Urine Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Draw (10cc) to determine eligibility (CBC, blood chemistries). Blood draw (20cc) at t=0 in fasting state for baseline measurement of biochemical markers (including carnitine, acylcarnitines, creatinine, and total lipid panel) Urine collection at t=0 Blood draw (20cc) at t=2 hours for measurement of biochemical markers (including carnitine, acylcarnitines, creatinine, and total lipid panel) Urine collection at t=2 hours Transformation of blood to establish lymphoblastoid cell lines (from blood samples collected at t=0 and t=2 hours)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Fasting: Other: Fasting blood and urine collection
  Interventions: Other: Fasting blood and urine collection

INTERVENTIONS:
Other: Fasting blood and urine collection — Not applicable no drugs dispensed

SUMMARY:
The current study is part of a large multi-investigator grant to look at the pharmacogenetics of a number of membrane transporters. Previously, the investigators have recruited a cohort of healthy volunteers (Studies of Pharmacogenetics in Ethnically-Diverse Populations, or SOPHIE) and have resequenced the coding region of a number of membrane transporter genes to identify genetic polymorphisms in these genes. Subjects in this cohort have agreed to be called back for recruitment in further studies based on their own genetic sequence, allowing the investigators the possibility to prospectively study the influence of genetic polymorphisms on particular phenotypes (i.e., genotype-to-phenotype studies). The investigators plan to take a genotype-to-phenotype approach to study the influence of specific polymorphisms in the novel organic cation transporter 2 (OCTN2) gene on carnitine and lipid metabolism in healthy subjects.

DETAILED DESCRIPTION:
Although OCTN2 is fairly well studied in its relationship with SCD, little is known about the carrier frequency of disease-causing alleles of OCTN2, or of more common functional polymorphisms in this gene. To address these issues, we screened for genetic variants in the OCTN2 coding region by direct sequencing of the exons and flanking intronic region of OCTN2 in a large sample (n = 276) of ethnically diverse subjects. In addition, we established lymphoblastoid cell lines from subjects homozygous for either allele of the previously identified promoter region variant, -207G>C. We found eight amino acid sequence variants of OCTN2, of which three (Phe17Leu, Leu144Phe, and Pro549Ser) were polymorphic in at least one ethnic group. When assayed for functional activity by expression in human embryonic kidney 293 cells, using as probes both the endogenous substrate (l-carnitine) and the organic cation tetraethylammonium, three variants showed functional differences from the reference OCTN2 (Phe17Leu, Tyr449Asp, Val481Phe; p < 0.05). Further studies of the Phe17Leu polymorphism showed a reduced V(max) for l-carnitine transport to approximately 50% of the reference OCTN2. Confocal microscopy studies using an OCTN2-GFP fusion protein showed that Phe17Leu had distinct subcellular localization from the reference OCTN2, with diffuse cytoplasmic retention of Phe17Leu, in contrast to reference OCTN2, which localized specifically to the plasma membrane. Lymphoblasts from subjects homozygous for the -207G allele showed increased l-carnitine transport compared with the -207C/C homozygotes (p < 0.05). This study suggests that although loss-of-function mutations in OCTN2 are likely to be rare, common variants of OCTN2 found in healthy populations may contribute to variation in the disposition of carnitine and some clinically used drugs.

ELIGIBILITY:
Inclusion Criteria:

* Previous participation in the "SOPHIE" study
* Between the ages of 18 and 40 years old
* Have a pre-selected genotype for OCTN1 and OCTN2
* Have been selected as healthy by medical history questionnaire and screening blood work (complete blood count [CBC], comprehensive metabolic panel).

Exclusion Criteria:

* Pregnant at the time of the study
* Have a new history indicating they are no longer healthy
* Taking a medication that could confound study results
* Individuals with anemia (hemoglobin < 12 g/dL), an elevation in liver enzymes to higher than double the respective normal value, or elevated creatinine concentrations (males ≥ 1.5 mg/dL, females ≥ 1.4 mg/dL).
* Do not consent to participate in the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy individuals per screening laboratory results and health questionnaire
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2005-01; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Giacomini, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States

REFERENCES:
- [Result] Urban TJ, Gallagher RC, Brown C, Castro RA, Lagpacan LL, Brett CM, Taylor TR, Carlson EJ, Ferrin TE, Burchard EG, Packman S, Giacomini KM. Functional genetic diversity in the high-affinity carnitine transporter OCTN2 (SLC22A5). Mol Pharmacol. 2006 Nov;70(5):1602-11. doi: 10.1124/mol.106.028126. Epub 2006 Aug 24. PMID 16931768